CLINICAL TRIAL: NCT05169450
Title: Efficacy of Diterpene Ginkgolides Meglumine Injection in Elderly Patients With Ischemic Stroke: A Post Hoc Analysis of a Randomized Controlled Trial
Brief Title: Efficacy of Diterpene Ginkgolides Meglumine Injection in Elderly Patients With Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ2013012
Record Dates: First submitted 2021-12-06; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Stroke; Ischemic Stroke; Nervous System Diseases; Cerebral Infarction; Brain Ischemia; Brain Infarction
Keywords: Diterpene Ginkgolides Meglumine Injection; acute ischemic stroke; effectiveness
MeSH Terms: conditions — Stroke; Ischemic Stroke; Nervous System Diseases; Cerebral Infarction; Brain Ischemia; Brain Infarction | interventions — ginaton

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diterpene ginkgolides meglumine injection (Experimental): The intervention group received daily single infusions of 25 mg diterpene ginkgolides meglumine injection (DGMI) diluted with 250 ml of 0.9% sodium chloride injection for 14 days.
  Interventions: Drug: Diterpene ginkgolides meglumine injection
- Ginaton (Active Comparator): The control group received once or twice a day infusion of 35-60mg Ginaton diluted with 250 ml of 0.9% sodium chloride injection for 14 days.
  Interventions: Drug: Ginaton

INTERVENTIONS:
Drug: Diterpene ginkgolides meglumine injection — Patients will receive intravenously administered diterpene ginkgolides meglumine injection, combined with guidelines-based standard care.
  Other Names: Ginkgolides Diterpene Lactone Meglumine Injection
  Arms: Diterpene ginkgolides meglumine injection
Drug: Ginaton — Patients will receive intravenously administered Ginaton, combined with guidelines-based standard care.
  Arms: Ginaton

SUMMARY:
A randomized positived-controlled study of Diterpene Ginkgolides Meglumine Injection (DGMI) vs Ginaton in patients with ischemic stroke (IS) was conducted between7/2013 and 4/2014. The study was designed to test efficacy of DGMI for IS. Post hoc analysis of this trial was conducted to evaluate the efficacy of DGMI in elderly (aged≥65 years) IS patients.

DETAILED DESCRIPTION:
To examine the efficacy of Diterpene Ginkgolides Meglumine Injection (DGMI) vs Ginaton in patients with ischemic stroke (IS) by age subgroups. The efficacy analysis was a post hoc analysis of data from a large randomized, controlled study was performed in a cohort of 998 IS patients. Patients were pooled and grouped by age (elderly aged ≥ 65 years and non-elderly aged < 65 years).Proportion of patients with Modified Rankin Scale (mRS) less than or equal to 1 at 90days is the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or older, and gender not limited;
* Between 2 and 4 weeks onset of ischemic stroke;
* The first onset, or always not obvious legacy of stroke sequela (mRS acuities were before the onset of 1);
* Understand and voluntarily signed informed consent.

Exclusion Criteria:

* Known severe liver or kidney dysfunction;
* Known allergies for ingredients in the investigational product;
* Known medical condition likely to limit survival to less than 3 months;
* Known dementia, mental impairment, or unsuitability for participation as judged by the investigators;
* Hemorrhage transformation after infarction, or bleeding tendency;
* Pregnancy or breastfeeding;
* Known lower extremity venous thrombosis;
* Having participated in others clinical trial within 1 month before randomization.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 998 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days
  Excellent functional outcome defined as an Modified Rankin Scale (mRS) score ≤ 1 at 90 days(scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death)

SECONDARY OUTCOMES:
Neurological deficit amelioration | 14 post-randomization days, 90days
  neurological deficit amelioration, which was defined as a change in the National Institutes of Health Stroke Scale (NIHSS) score (range = 0-42, with higher scores indicating more severe strokes) from baseline to D14
Patient quality of life | 14 post-randomization days, 90days
  Patient quality of life, as measured using the EuroQol questionnaire [consisting of two parts: EuroQol-5 Dimension(EQ-5D) and EQ visual analog scale (EQ-VAS)]. A value of 100 on this scale indicates a perfect score for health, whereas a score of 0 indicates death. The EQ-5D index score is measured on a scale of 0 (death) to 1 (full health).

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Resource links provided by the National Library of Medicine — https://druginfo.nlm.nih.gov/drugportal/name/Meglumine
- See also: Resource links provided by the National Library of Medicine — https://druginfo.nlm.nih.gov/drugportal/name/Ginkgo+biloba